CLINICAL TRIAL: NCT02217059
Title: Congruence of Emergency Department Attendings' Predictions of Hypertension With Results of Home Blood Pressure Monitoring
Brief Title: Emergency Department Home Blood Pressure Monitoring and BpTRU Study
Status: Completed | Type: Observational
Sponsor: Rhode Island Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: UEMF0000
Record Dates: First submitted 2014-08-07; First posted 2014-08-15 (Estimated); Last update posted 2017-11-29 (Actual); Status verified 2016-03

CONDITIONS: Hypertension
Keywords: Emergency Medical Services; Emergency Care; Hypertension; BpTRU; Blood pressure
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Prehypertension: Using the JNC7 definition
- Stage I Hypertension: Using the JNC7 definition
- Stage II Hypertension: Using the JNC7 definition

SUMMARY:
The purpose of this study is to evaluate the Congruence of Emergency Department (ED) Attendings' Predictions of Hypertension with Results of Home Blood Pressure Monitoring.

DETAILED DESCRIPTION:
Evaluate the Congruence of Emergency Department (ED) Attendings' Predictions of Hypertension with Results of Home Blood Pressure Monitoring & evaluate reliability of ED measured elevated blood pressure compared to the BpTRU

ELIGIBILITY:
Inclusion Criteria:

* One elevated blood pressure greater than 120 systolic and/or 80 diastolic
* BpTRU device blood pressure greater than 120 systolic and/or 80 diastolic while in ED

Exclusion Criteria:

* Prior history of hypertension
* Currently on antihypertensives or receiving prescription on discharge
* Pregnancy
* History of atrial fibrillation
* Dialysis patient
* Nursing home or rehabilitation center resident
* Admitted
* Moving out of the area in next 30 days
* Substance abuse
* Prisoner
* Presenting for psychiatric complaint requiring constant observation
* Inability to give informed consent (intoxicated, altered, non-English speaking)
* Presenting with symptoms of hypertensive emergency
* Inability to demonstrate adequate use of the home blood pressure device in the ED
* Arm circumference less than 9 inches or greater than 17 inches

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Emergency Department
Sampling Method: Probability Sample
Enrollment: 105 (Actual)
Dates: Start 2014-08; Primary Completion 2017-07 (Actual); Study Completion 2017-07 (Actual)

PRIMARY OUTCOMES:
The percentage of emergency department attendings that accurately predict which patients meet criteria for hypertension in two week follow-up using home blood pressure monitoring. | 18 months

SECONDARY OUTCOMES:
The predictive value of the emergency department measured blood pressure by the standard ED blood pressure device, BpTRU device, and home blood pressure device for hypertension in follow-up | 18 months

CONTACTS AND LOCATIONS:
Locations (1):
- Rhode Island Hospital, Providence, Rhode Island, United States

IPD SHARING:
Plan to Share IPD: No